CLINICAL TRIAL: NCT03392753
Title: Randomised Controlled Trial of Mechanochemical Ablation Versus Cyanoacrylate Adhesive for the Treatment of Varicose Veins
Brief Title: Mechanochemical Ablation Compared to Cyanoacrylate Adhesive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17/LO/1457
Record Dates: First submitted 2017-11-28; First posted 2018-01-08 (Actual); Results first posted 2021-12-07 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins | interventions — MK 6 cyanoacrylate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: An internet-based randomisation service will be used Outcome assessors will be blinded as to treatment offered
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanochemical ablation (MOCA) (Active Comparator): Mechanochemical ablation using the ClariVein® mechanochemical ablation (MOCA) device (Vascular Insights, Madison, CT, USA).
  Interventions: Procedure: Mechanochemical ablation
- Cyanoacrylate adhesive (CAE) (Active Comparator): Cyanoacrylate using the VenaSealTM Closure System (Medtronic, Minneapolis, Minnesota, USA).
  Interventions: Procedure: Cyanoacrylate adhesive

INTERVENTIONS:
Procedure: Mechanochemical ablation — Treatment of incompetent saphenous veins using mechanochemical ablation (Clarivein)
  Arms: Mechanochemical ablation (MOCA)
Procedure: Cyanoacrylate adhesive — Treatment of incompetent saphenous veins using cyanoacrylate (VenaSealTM)
  Arms: Cyanoacrylate adhesive (CAE)

SUMMARY:
This study will be comparing the treatment of varicose veins using either mechanochemical ablation (MOCA) or cyanoacrylate adhesive (CAE). Patients will be randomised to receiving either MOCA or CAE.

The pain scores, clinical scores, quality of life scores, occlusion and re-intervention rate at 2 weeks, 3, 6 and 12 months as well as the cost effectiveness of each intervention will be assessed.

DETAILED DESCRIPTION:
This will be a randomised clinical trial comparing MOCA to CAE. Patients will be randomised into group A (MOCA) or group B (CAE). Only the endovenous ablation part of the procedure will be randomised while the decision as to whether patients should receive treatment of their varicose tributaries will be at the discretion of the clinical team.

The device used for MOCA (group A) will be the ClariVein® mechanochemical ablation (MOCA) device (Vascular Insights, Madison, CT, USA).

The device used for CAE (group B) will be the VenaSealTM Closure System (Medtronic, Minneapolis, Minnesota, USA).

Re-intervention of the treated saphenous veins will not be decided until at least 3 months after their initial procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Symptomatic GSV or SSV vein reflux > 0.5 seconds on colour Duplex

Exclusion Criteria:

* Current DVT
* Recurrent varicose veins
* Arterial disease (ABPI<0.8)
* Vein diameter < 3mm
* Patient who are unwilling to participate
* Inability or unwillingness to complete questionnaires
* Adverse reaction to sclerosant or cyanoacrylate
* Not been involved in another venous trial for at least 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alun H Davies, Principal Investigator — Imperial College London
Locations (1):
- Charing Cross Hospital, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belramman A, Bootun R, Tang TY, Lane TRA, Davies AH. Pain Outcomes Following Mechanochemical Ablation vs Cyanoacrylate Adhesive for the Treatment of Primary Truncal Saphenous Vein Incompetence: The MOCCA Randomized Clinical Trial. JAMA Surg. 2022 May 1;157(5):395-404. doi: 10.1001/jamasurg.2022.0298. PMID 35385061
- [Derived] Belramman A, Bootun R, Tang TY, Lane TRA, Davies AH. Mechanochemical ablation versus cyanoacrylate adhesive for the treatment of varicose veins: study protocol for a randomised controlled trial. Trials. 2018 Aug 7;19(1):428. doi: 10.1186/s13063-018-2807-0. PMID 30086774

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 2017 and February 2020
  Recruitment location:
  1. Charing Cross Hospital (Imperial College Healthcare NHS Trust) in London, UK;
  2. Singapore General Hospital;
  3. Sengkang General Hospital (Singapore)
Pre-assignment Details: 167 patients recruited
Period: Overall Study
Arm/Group | Mechanochemical Ablation (MOCA) | Cyanoacrylate Adhesive (CAE)
Started | 83 | 84
Completed | 47 | 50
Not Completed | 36 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mechanochemical Ablation (MOCA) | Cyanoacrylate Adhesive (CAE) | Total
Number analyzed (Participants) | 83 | 84 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (16) | 55 (15) | 56 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 46 | 99
  Male | 30 | 38 | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 50 | 50 | 100
  Singapore | 33 | 34 | 67

OUTCOME MEASURES:

1. Primary Outcome: Pain Score During Ablation
Description: Pain score during saphenous vein ablation using a 0-100mm visual analogue scale (0=no pain; 100=worst pain)
Time Frame: On day 0 immediately following vein ablation
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Mechanochemical Ablation (MOCA) | Cyanoacrylate Adhesive (CAE)
Number analyzed (Participants) | 83 | 84
Units on a scale | 24 [24 to 44.7] | 20 [9 to 42]

2. Secondary Outcome: Pain Score at the End of the Procedure
Description: Pain score at the end of the procedure using a 0-100mm visual analogue scale (0=no pain; 100=worst pain)
Time Frame: On day 0 following vein ablation and any tributary treatment
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Mechanochemical Ablation (MOCA) | Cyanoacrylate Adhesive (CAE)
Number analyzed (Participants) | 83 | 84
Units on a scale | 8 [3 to 22] | 11 [4 to 27]

3. Secondary Outcome: Generic Quality of Life as Per EQ-5D Questionnaire
Description: Using the EuroQoL's EQ-5D questionnaire (-0.085=worse quality of life; 1.000=best quality of life)
Time Frame: Recorded at 12 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Mechanochemical Ablation (MOCA) | Cyanoacrylate Adhesive (CAE)
Number analyzed (Participants) | 47 | 50
score on a scale | 1 [0.74 to 1] | 1 [0.73 to 1]

4. Secondary Outcome: Disease Specific Quality of Life as Per the AVVQ
Description: Using the Aberdeen Varicose Vein Questionnaire (AVVQ) questionnaire (0=best quality of life; 100=worse quality of life)
Time Frame: Recorded at 12 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Mechanochemical Ablation (MOCA) | Cyanoacrylate Adhesive (CAE)
Number analyzed (Participants) | 47 | 50
score on a scale | 4 [0 to 11.9] | 5.9 [1.4 to 13.4]

5. Secondary Outcome: Disease Specific Quality of Life as Per the CIVIQ-20
Description: Using the CIVIQ-20 questionnaire (0=best quality of life; 100=worse quality of life)
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Mechanochemical Ablation (MOCA) | Cyanoacrylate Adhesive (CAE)
Number analyzed (Participants) | 47 | 50
score on a scale | 3.5 [0 to 20] | 7.1 [0.75 to 21.4]

6. Secondary Outcome: Clinical Change as Per VCSS
Description: Using the Venous Clinical Severity Score (VCSS) (0=best; 30=worse)
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Mechanochemical Ablation (MOCA) | Cyanoacrylate Adhesive (CAE)
Number analyzed (Participants) | 47 | 50
score on a scale | 2 [1 to 3] | 2 [1 to 3]

7. Secondary Outcome: Pain Score Over the First 10 Days
Description: Pain score over the first 10 days using a 0-100mm visual analogue scale (0=no pain; 100=worst pain). The mean pain score was recorded daily and a mean value was calculated.
Time Frame: For the first 10 days since procedure
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Mechanochemical Ablation (MOCA) | Cyanoacrylate Adhesive (CAE)
Number analyzed (Participants) | 47 | 50
Units on a scale | 10.5 [3 to 16] | 7 [2.5 to 19]

8. Secondary Outcome: Degree of Bruising at 2 Weeks
Description: Degree of bruising at 2 weeks using a categorical 0-5 bruising scale (0=no bruising; 5=bruising extending beyond treated segment). The outcome measured is the number of participants with a degree of bruising between category 0-1.
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Mechanochemical Ablation (MOCA) | Cyanoacrylate Adhesive (CAE)
Number analyzed (Participants) | 59 | 71
participants | 53 | 59

9. Secondary Outcome: Time to Return to Normal Activities
Description: Length of time in days until normal activities are resumed
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Mechanochemical Ablation (MOCA) | Cyanoacrylate Adhesive (CAE)
Number analyzed (Participants) | 71 | 77
days | 7 [4 to 10] | 8.5 [4 to 10]

10. Secondary Outcome: Occlusion Rates
Description: Rate of occlusion as assessed by duplex ultrasound
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mechanochemical Ablation (MOCA) | Cyanoacrylate Adhesive (CAE)
Number analyzed (Participants) | 33 | 34
Participants | 29 | 31

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Mechanochemical Ablation (MOCA) | Cyanoacrylate Adhesive (CAE)
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/84
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/84
Other Adverse Events (participants affected / at risk) | 0/83 | 2/84
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mechanochemical Ablation (MOCA) (N=83) | Cyanoacrylate Adhesive (CAE) (N=84)
Phlebitis (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT03392753/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT03392753/SAP_001.pdf